CLINICAL TRIAL: NCT05750992
Title: Ultrasound Guided Transversus Abdominis Plane Block (TAPB) vs Surgical TAPB With Bupivacaine for Acute Pain Control in Cesarean Section: A Randomized Clinical Trial
Brief Title: Ultrasound Guided TAPB vs Surgical TAPB With Bupivacaine in Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFM-IRB 00012367- 23-02-006
Record Dates: First submitted 2023-02-19; First posted 2023-03-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Cesarean Section; Ultrasound Guided Transversus Abdominis Plane Block; Surgical Transversus Abdominis Plane Block; Bupivacaine; Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Saline Solution; Fentanyl; Meperidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical TAP block (Active Comparator): twenty-five pregnant women will receive surgical TAP block performed by 40 ml of 0.25% bupivacaine (10 ml 0.5% bupivacaine bilaterally diluted with 10cc normal saline and 100 μg of fentanyl), the total volume was divided equally and administered bilaterally by the surgeon.
  Interventions: Procedure: surgical TAP block
- US guided TAP block (Active Comparator): 25 pregnant women will receive US guided T.A.P block performed by 40 ml of 0.25% bupivacaine (10 ml 0.5% bupivacaine bilaterally diluted with 10cc normal saline and 100 μg of fentanyl), the total volume was divided equally and administered bilaterally.
  Interventions: Procedure: US guided TAP block

INTERVENTIONS:
Procedure: surgical TAP block — performed by 40 ml of 0.25% bupivacaine (10 ml 0.5% bupivacaine bilaterally diluted with 10cc normal saline and 100 μg of fentanyl), the total volume was divided equally and administered bilaterally by the surgeon.
  Other Names: bupivacaine, normal saline, fentanyl, pethidine
  Arms: surgical TAP block
Procedure: US guided TAP block — performed by 40 ml of 0.25% bupivacaine (10 ml 0.5% bupivacaine bilaterally diluted with 10cc normal saline and 100 μg of fentanyl), the total volume was divided equally and administered bilaterally.
  Other Names: bupivacaine, normal saline, fentanyl , pethidine
  Arms: US guided TAP block

SUMMARY:
The aim of this study is to compare Surgical Transversus abdominis plane block and Ultrasound guided transversus abdominis plane block (TAPB) as a postoperative analgesic regimen in female patients undergoing elective cesarean delivery.

DETAILED DESCRIPTION:
Caesarean delivery rates have been increasing worldwide nowadays. At rate of [52%], Egypt stands out among countries with the world's highest cesarean delivery percentages . Within the Arab region, rate of cesarean section far higher in Egypt than other Arab countries.

A much simpler and theoretically superior means of establishing a TAP block. When using a transcutaneous (conventional) approach there is always the risk of peritoneal puncture with its attendant complications. Moreover, there are technical difficulties, especially in obese women and the procedure requires specialist equipment, a skilled operator and training in ultrasonography. Our approach obviates these risks and difficulties because the procedure is carried out under direct vision, and it is much easier to perform by the surgeon during caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Full term pregnant women
* Older than 21 years of age
* Had elective cesarean section with Pfannenstiel incision.

Exclusion Criteria:

* Patients with cesarean section using different surgical incision
* History of addiction [including opioids and benzodiazepines]
* Allergy to the anesthetic analgesia
* Psychological disorders
* Coagulopathies
* Infection at the block injection site.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to perform block. | 1 hour postoperatively
  The time taken to perform the block will be recorded by an independent observer.

SECONDARY OUTCOMES:
Heart rate | 24 hours postoperatively
  Patients hemodynamics (heart rate will be recorded)
Mean arterial blood pressure | 24 hours postoperatively
  Patients hemodynamics (mean arterial blood pressure will be recorded)
Pain score | 24 hours postoperatively
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Time to first analgesic request | 24 hours postoperatively
  The time to first analgesic request will be recorded
Amount of post operative analgesic consumption | 24 hours postoperatively
  The amount of post operative analgesic consumption will be recorded
Time spent in operating room | 24 hours postoperatively
  The time spent in operating room will be recorded
Incidence of Adverse reactions | 24 hours postoperatively
  Adverse events will be recorded such as nausea, vomiting, hypotension (Mean arterial blood pressure < 20% of baseline readings and will be managed by ephedrine 5 mg IV and/or normal saline IV) and bradycardia (heart rate < 60 beats/min and will be managed by atropine 0.6 mg IV).

CONTACTS AND LOCATIONS:
Locations (1):
- Kohaf, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principle investigator
Supporting Information: Study Protocol, SAP
Time Frame: for one year after completion of the study